CLINICAL TRIAL: NCT01471509
Title: The Effect of Ingestion of Foods on the Plasma Glucose and Insulin Response in Subjects With Type 2 Diabetes: Protein, Amino Acids & Insulin & Glucagon Secretion in Humans
Brief Title: Protein, Amino Acids & Insulin & Glucagon Secretion in Humans
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frank Q. Nuttall, MD, PhD, Section of Endocrinology, Metabolism & Nutrition, Professor of Medicine, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 676
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome
Keywords: Glycemic Index; LoBAG Diet; Insulin; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Insulin Resistance | interventions — Water; Glucose; Amino Acids; Food

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): 240 ml water
  Interventions: Other: water, glucose with or without amino acid
- glucose (Active Comparator): 50 g glucose
  Interventions: Other: water, glucose with or without amino acid
- Amino acid (Active Comparator): 1 mmol amino acid/kg lean body mass
  Interventions: Other: water, glucose with or without amino acid
- amino acid plus glucose (Active Comparator): 50 g glucose plus 1 mmol amino acid/kg lean body mass
  Interventions: Other: water, glucose with or without amino acid

INTERVENTIONS:
Other: water, glucose with or without amino acid — 240 ml water, 50 g glucose ± 1 mmol amino acid/kg lean body mass
  Other Names: foods or food constituents

SUMMARY:
The purpose of this study is to determine the effect of various foods and/or food substances such as fats or proteins on the blood glucose and insulin concentrations in people with and without type 2 diabetes.

DETAILED DESCRIPTION:
Various foods or food substances are given as a test meal. The metabolic response is determined at various times after the administration of the meal (e.g. blood glucose, and other hormones and metabolites).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with or without type 2 diabetes
* C-Peptide > 1.5 ng/ml
* Able to come to the Minneapolis VA Medical Center on several occasions over 2-4 weeks

Exclusion Criteria:

* Body mass index > 40
* hematologic abnormalities
* liver disease
* kidney disease
* congestive heart failure
* life threatening malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1982-08; Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose concentration | several time points after ingestion of test substance
  Test substances will be given at 0800 hr and blood drawn at several time points up to 5 hours after the meal.

SECONDARY OUTCOMES:
Change in serum insulin concentration | Several time points after ingestion of test substance
  Test substances will be given at 0800 hr and blood drawn at several time points up to 5 hours after the meal.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Q Nuttall, M.D., Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Iverson JF, Gannon MC, Nuttall FQ. Ingestion of leucine + phenylalanine with glucose produces an additive effect on serum insulin but less than additive effect on plasma glucose. J Amino Acids. 2013;2013:964637. doi: 10.1155/2013/964637. Epub 2013 Jul 29. PMID 23984046
- [Background] Iverson JF, Gannon MC, Nuttall FQ. Interaction of ingested leucine with glycine on insulin and glucose concentrations. J Amino Acids. 2014;2014:521941. doi: 10.1155/2014/521941. Epub 2014 Jul 10. PMID 25120925
- [Result] Nuttall FQ, Mooradian AD, Gannon MC, Billington C, Krezowski P. Effect of protein ingestion on the glucose and insulin response to a standardized oral glucose load. Diabetes Care. 1984 Sep-Oct;7(5):465-70. doi: 10.2337/diacare.7.5.465. PMID 6389060
- [Result] Nuttall FQ, Gannon MC, Wald JL, Ahmed M. Plasma glucose and insulin profiles in normal subjects ingesting diets of varying carbohydrate, fat, and protein content. J Am Coll Nutr. 1985;4(4):437-50. doi: 10.1080/07315724.1985.10720086. PMID 3900180
- [Result] Krezowski PA, Nuttall FQ, Gannon MC, Bartosh NH. The effect of protein ingestion on the metabolic response to oral glucose in normal individuals. Am J Clin Nutr. 1986 Dec;44(6):847-56. doi: 10.1093/ajcn/44.6.847. PMID 3538843
- [Result] Gannon MC, Nuttall FQ, Krezowski PA, Billington CJ, Parker S. The serum insulin and plasma glucose responses to milk and fruit products in type 2 (non-insulin-dependent) diabetic patients. Diabetologia. 1986 Nov;29(11):784-91. doi: 10.1007/BF00873217. PMID 3545955
- [Result] Krezowski PA, Nuttall FQ, Gannon MC, Billington CJ, Parker S. Insulin and glucose responses to various starch-containing foods in type II diabetic subjects. Diabetes Care. 1987 Mar-Apr;10(2):205-12. doi: 10.2337/diacare.10.2.205. PMID 3556106
- [Result] Gannon MC, Nuttall FQ. Factors affecting interpretation of postprandial glucose and insulin areas. Diabetes Care. 1987 Nov-Dec;10(6):759-63. doi: 10.2337/diacare.10.6.759. PMID 3322731
- [Result] Nuttall FQ, Gannon MC. Quantitative importance of dietary constituents other than glucose as insulin secretagogues in type II diabetes. Diabetes Care. 1988 Jan;11(1):72-6. doi: 10.2337/diacare.11.1.72. PMID 3276480
- [Result] Gannon MC, Nuttall FQ, Neil BJ, Westphal SA. The insulin and glucose responses to meals of glucose plus various proteins in type II diabetic subjects. Metabolism. 1988 Nov;37(11):1081-8. doi: 10.1016/0026-0495(88)90072-8. PMID 3054432
- [Result] Gannon MC, Nuttall FQ, Westphal SA, Neil BJ, Seaquist ER. Effects of dose of ingested glucose on plasma metabolite and hormone responses in type II diabetic subjects. Diabetes Care. 1989 Sep;12(8):544-52. doi: 10.2337/diacare.12.8.544. PMID 2673694
- [Result] Nuttall FQ, Gannon MC. Metabolic response to egg white and cottage cheese protein in normal subjects. Metabolism. 1990 Jul;39(7):749-55. doi: 10.1016/0026-0495(90)90112-p. PMID 2195298
- [Result] Westphal SA, Gannon MC, Nuttall FQ. Metabolic response to glucose ingested with various amounts of protein. Am J Clin Nutr. 1990 Aug;52(2):267-72. doi: 10.1093/ajcn/52.2.267. PMID 2197851
- [Result] Gannon MC, Nuttall FQ. Quantitation of the glucose area response to a meal. Diabetes Care. 1990 Oct;13(10):1095-6. doi: 10.2337/diacare.13.10.1095a. No abstract available. PMID 2209312
- [Result] Nuttall FQ, Gannon MC. Plasma glucose and insulin response to macronutrients in nondiabetic and NIDDM subjects. Diabetes Care. 1991 Sep;14(9):824-38. doi: 10.2337/diacare.14.9.824. PMID 1959475
- [Result] Nuttall FQ, Gannon MC, Burmeister LA, Lane JT, Pyzdrowski KL. The metabolic response to various doses of fructose in type II diabetic subjects. Metabolism. 1992 May;41(5):510-7. doi: 10.1016/0026-0495(92)90210-2. PMID 1588830
- [Result] Gannon MC, Nuttall FQ, Lane JT, Burmeister LA. Metabolic response to cottage cheese or egg white protein, with or without glucose, in type II diabetic subjects. Metabolism. 1992 Oct;41(10):1137-45. doi: 10.1016/0026-0495(92)90300-y. PMID 1406301
- [Result] Khan MA, Gannon MC, Nuttall FQ. Glucose appearance rate following protein ingestion in normal subjects. J Am Coll Nutr. 1992 Dec;11(6):701-6. doi: 10.1080/07315724.1992.10718270. PMID 1460185
- [Result] Gannon MC, Ercan N, Westphal SA, Nuttall FQ. Effect of added fat on plasma glucose and insulin response to ingested potato in individuals with NIDDM. Diabetes Care. 1993 Jun;16(6):874-80. doi: 10.2337/diacare.16.6.874. PMID 8325201
- [Result] Ercan N, Nuttall FQ, Gannon MC, Lane JT, Burmeister LA, Westphal SA. Plasma glucose and insulin responses to bananas of varying ripeness in persons with noninsulin-dependent diabetes mellitus. J Am Coll Nutr. 1993 Dec;12(6):703-9. doi: 10.1080/07315724.1993.10718362. PMID 8294726
- [Result] Ercan N, Nuttall FQ, Gannon MC, Redmon JB, Sheridan KJ. Effects of glucose, galactose, and lactose ingestion on the plasma glucose and insulin response in persons with non-insulin-dependent diabetes mellitus. Metabolism. 1993 Dec;42(12):1560-7. doi: 10.1016/0026-0495(93)90151-d. PMID 8246770
- [Result] Ercan N, Gannon MC, Nuttall FQ. Effect of added fat on the plasma glucose and insulin response to ingested potato given in various combinations as two meals in normal individuals. Diabetes Care. 1994 Dec;17(12):1453-9. doi: 10.2337/diacare.17.12.1453. PMID 7882816
- [Result] Gannon MC, Nuttall FQ, Lane JT, Fang S, Gupta V, Sandhofer CR. Effect of 24 hours of starvation on plasma glucose and insulin concentrations in subjects with untreated non-insulin-dependent diabetes mellitus. Metabolism. 1996 Apr;45(4):492-7. doi: 10.1016/s0026-0495(96)90225-5. PMID 8609837
- [Result] Gannon MC, Nuttall FQ, Grant CT, Ercan-Fang S, Ercan-Fang N. Stimulation of insulin secretion by fructose ingested with protein in people with untreated type 2 diabetes. Diabetes Care. 1998 Jan;21(1):16-22. doi: 10.2337/diacare.21.1.16. PMID 9538964
- [Result] Holtschlag DJ, Gannon MC, Nuttall FQ. State-space models of insulin and glucose responses to diets of varying nutrient content in men and women. J Appl Physiol (1985). 1998 Sep;85(3):935-45. doi: 10.1152/jappl.1998.85.3.935. PMID 9729567
- [Result] Gannon MC, Nuttall FQ, Westphal SA, Fang S, Ercan-Fang N. Acute metabolic response to high-carbohydrate, high-starch meals compared with moderate-carbohydrate, low-starch meals in subjects with type 2 diabetes. Diabetes Care. 1998 Oct;21(10):1619-26. doi: 10.2337/diacare.21.10.1619. PMID 9773720
- [Result] Nuttall FQ, Khan MA, Gannon MC. Peripheral glucose appearance rate following fructose ingestion in normal subjects. Metabolism. 2000 Dec;49(12):1565-71. doi: 10.1053/meta.2000.18553. PMID 11145118
- [Result] Gannon MC, Khan MA, Nuttall FQ. Glucose appearance rate after the ingestion of galactose. Metabolism. 2001 Jan;50(1):93-8. doi: 10.1053/meta.2001.19442. PMID 11172481
- [Result] Gannon MC, Nuttall JA, Damberg G, Gupta V, Nuttall FQ. Effect of protein ingestion on the glucose appearance rate in people with type 2 diabetes. J Clin Endocrinol Metab. 2001 Mar;86(3):1040-7. doi: 10.1210/jcem.86.3.7263. PMID 11238483
- [Result] Saeed A, Jones SA, Nuttall FQ, Gannon MC. A fasting-induced decrease in plasma glucose concentration does not affect the insulin response to ingested protein in people with type 2 diabetes. Metabolism. 2002 Aug;51(8):1027-33. doi: 10.1053/meta.2002.34033. PMID 12145777
- [Result] Gannon MC, Nuttall JA, Nuttall FQ. Oral arginine does not stimulate an increase in insulin concentration but delays glucose disposal. Am J Clin Nutr. 2002 Nov;76(5):1016-22. doi: 10.1093/ajcn/76.5.1016. PMID 12399273
- [Result] Gannon MC, Nuttall JA, Nuttall FQ. The metabolic response to ingested glycine. Am J Clin Nutr. 2002 Dec;76(6):1302-7. doi: 10.1093/ajcn/76.6.1302. PMID 12450897
- [Result] Nuttall FQ, Gannon MC, Saeed A, Jordan K, Hoover H. The metabolic response of subjects with type 2 diabetes to a high-protein, weight-maintenance diet. J Clin Endocrinol Metab. 2003 Aug;88(8):3577-83. doi: 10.1210/jc.2003-030419. PMID 12915639
- [Result] Gannon MC, Nuttall FQ, Saeed A, Jordan K, Hoover H. An increase in dietary protein improves the blood glucose response in persons with type 2 diabetes. Am J Clin Nutr. 2003 Oct;78(4):734-41. doi: 10.1093/ajcn/78.4.734. PMID 14522731
- [Result] Nuttall FQ, Gannon MC, Jordan K. The metabolic response to ingestion of proline with and without glucose. Metabolism. 2004 Feb;53(2):241-6. doi: 10.1016/j.metabol.2003.09.013. PMID 14767878
- [Result] Gannon MC, Nuttall FQ. Effect of a high-protein, low-carbohydrate diet on blood glucose control in people with type 2 diabetes. Diabetes. 2004 Sep;53(9):2375-82. doi: 10.2337/diabetes.53.9.2375. PMID 15331548
- [Result] Nuttall FQ, Gannon MC. The metabolic response to a high-protein, low-carbohydrate diet in men with type 2 diabetes mellitus. Metabolism. 2006 Feb;55(2):243-51. doi: 10.1016/j.metabol.2005.08.027. PMID 16423633
- [Result] Nuttall FQ, Schweim KJ, Gannon MC. Effect of orally administered phenylalanine with and without glucose on insulin, glucagon and glucose concentrations. Horm Metab Res. 2006 Aug;38(8):518-23. doi: 10.1055/s-2006-949523. PMID 16941278
- [Result] Kalogeropoulou D, Lafave L, Schweim K, Gannon MC, Nuttall FQ. Leucine, when ingested with glucose, synergistically stimulates insulin secretion and lowers blood glucose. Metabolism. 2008 Dec;57(12):1747-52. doi: 10.1016/j.metabol.2008.09.001. PMID 19013300
- [Result] Kalogeropoulou D, LaFave L, Schweim K, Gannon MC, Nuttall FQ. Lysine ingestion markedly attenuates the glucose response to ingested glucose without a change in insulin response. Am J Clin Nutr. 2009 Aug;90(2):314-20. doi: 10.3945/ajcn.2008.27381. Epub 2009 Jun 24. PMID 19553295
- [Result] Radulescu A, Hassan Y, Gannon MC, Nuttall FQ. The degree of saturation of fatty acids in dietary fats does not affect the metabolic response to ingested carbohydrate. J Am Coll Nutr. 2009 Jun;28(3):286-95. doi: 10.1080/07315724.2009.10719783. PMID 20150602
- [Result] Radulescu A, Gannon MC, Nuttall FQ. The effect on glucagon, glucagon-like peptide-1, total and acyl-ghrelin of dietary fats ingested with and without potato. J Clin Endocrinol Metab. 2010 Jul;95(7):3385-91. doi: 10.1210/jc.2009-2559. Epub 2010 May 5. PMID 20444922
- [Result] Gannon MC, Nuttall FQ. Amino acid ingestion and glucose metabolism--a review. IUBMB Life. 2010 Sep;62(9):660-8. doi: 10.1002/iub.375. PMID 20882645